CLINICAL TRIAL: NCT03946137
Title: Chest Therapy and Postural Control in Children With Crhonic Neurological Patology
Brief Title: Chest Therapy and Postural Education in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Moreno Bermejo, Physiotherapist, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Complutense University
Record Dates: First submitted 2019-04-23; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Neurologic Disorder; Respiratory Complication; Child
Keywords: Neurological chronic disorder; Child; Chest therapy; Educational intervention; Postural hygiene
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Multicentric experimental study before-after with intervention of Chest physiotherapy and workshops of postural hygiene in 30 children from 0 to 6 years with chronic neurological diseases and respiratory complications.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sample (Experimental): 30 patients of both sexes aged between 0 and 6 years with chronic neurological involvement with respiratory complications.
  Individual sessions of chest therapy every fifteen days for three months, in total 6 respiratory physiotherapy sessions of 30 minutes each were performed. And the postural hygiene workshops were given to the parents, this educational intervention was carried out at the beginning of the study, at 3 months and at 6 months from the beginning. Each intervention lasted 4 hours with theoretical and practical part.
  Interventions: Other: Chest Therapy; Other: Postural Hygiene

INTERVENTIONS:
Other: Chest Therapy — The sessions of chest therapy were based on airway clearance techniques (hyper manual insufflations, abdominal thoracic compressions and manually assisted cough)
  Other Names: Airways clearance techniques
Other: Postural Hygiene — Postural hygiene workshops were taught through a theoretical presentation with the help of slides and practical exercises in small groups (2-4 parents per group).
  Other Names: Postural hygiene workshop

SUMMARY:
INTRODUCTION: Neurological Chronic disease leads to motor disability and associated pathologies. Numerous studies agree that the lack of prevention and treatment in pulmonary health in children with disabilities results in increased morbidity and mortality, increased medical care and costs in care, and, for patients and their caregivers, decrease in their quality of life OBJECTIVE: The objective of this study is to assess if children with chronic neurological disease and respiratory disease benefit from airway clearance techniques and postural hygiene workshops to optimize their respiratory status and quality of life. PATIENTS AND METHODS: Multicenter experimental study before-after with intervention of chest therapy and workshops of postural hygiene in 30 children from 0 to 6 years with chronic neurological affectation and respiratory complications. Respiratory clinical variables, volume of expectorated secretions, PedsQL pediatric quality of life questionnaires were evaluated and the number of exacerbations due to respiratory complications was recorded.

DETAILED DESCRIPTION:
There are few studies that apply and evaluate respiratory physiotherapy and / or postural hygiene in children with neurological affections. This study aims to improve the quality and effectiveness of physiotherapy interventions in paediatric patients with neurological problems and respiratory symptomatology, providing scientific evidence to respiratory physiotherapy protocols that are carried out in daily clinical practice and implementing the practice of therapeutic education on postural hygiene.

HYPOTHESIS: Children with neurological chronic disease and respiratory affection benefit from mucociliary clearance techniques and workshops on postural hygiene to optimize respiratory status and quality of life.

OBJECTIVES

* To evaluate the effectiveness of mucociliary clearance techniques in improving respiratory clinical signs and to increase expectoration of bronchial secretions in children with chronic neurological disease.
* To analyse the effectiveness of mucociliary clearance techniques combined with workshops to improve the quality of life of children with chronic neurological disease with respiratory complications.
* Establish the effectiveness of mucociliary clearance techniques and workshops to reduce the number of exacerbations due to respiratory infection in children with chronic neurological disease.
* To determine the effectiveness of mucociliary clearance techniques and workshops to reduce hospital admissions for respiratory complications in children with chronic neurological disease.
* MATERIAL AND METHODS It is an experimental study before - after a single group of children with non-progressive chronic neurological affectation (Cerebral Palsy, Down Syndrome, encephalopathies, ...) and respiratory involvement with intervention of chest therapy and workshops of postural hygiene directed to their parents or guardians Each individual has been their own control in the successive evaluations. The physiotherapist who has performed the techniques of chest therapy and workshops has been the same as the physiotherapist evaluator, so that there has been neither simple nor double blind.

The project was previously approved by the Clinical Research Ethics Committee of the San Carlos Clinical University Hospital (internal code nº 15/152-E); He was awarded the 2014 Research Fellowship of the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR).

ESTIMATION OF SAMPLE SIZE The sample size necessary to obtain a good internal validity was calculated, considering a normal distribution of the data, making a population estimate according to Granmo for paired means (repeated in a group). And the Bonferroni correction was taken into account, that is, the significance of at least 0.05 divided by the number of comparisons (in this case 8) was considered for each contrast.

So, estimating a significance of 0.00625 (0.05 / 8) and a power of 0.8, in a bilateral contrast, 27 subjects are required to detect a difference equal to or greater than 3.5 units. A standard deviation of 5 is assumed.

The participants were recruited from four centres of early care and foundations of the Community of Madrid. From their respective centres, all the parents of children with chronic neurological syndromes, who could enter the study according to the inclusion and exclusion criteria previously described, participated in the project.

The informed consent of the parents or guardians of each participant was filed outside their medical history and they were informed of the confidentiality of the data according to the Organic Law 15/99 of December 13 of Data Protection of personal character.

Subsequently, a first evaluation of the participants was performed, in which the descriptive data, the clinical exams, the number of exacerbations that each participant underwent during the 6 months prior to the beginning of the study were collected and the PedsQL quality of life questionnaires Through a personal interview with the parents.

After this first evaluation, the clinical evaluations were performed, including the clinical exams of the participants before and after each session. And, after each session, the volume of secretions expectorated by each participant was measured. In the last session (session 6) the PedsQL quality of life questionnaires were completed again.

Finally, in the evaluation of evolutionary control, clinical examinations were performed, the PedsQL quality of life questionnaires were again completed and the number of exacerbations due to respiratory complications that each participant had during the six months after the study was started.

Chest therapy was performed twice a month. The intervention of the workshops was done every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose parents or guardians have signed informed consent.
* Patients of both sexes whose ages are between 0 and 6 years.
* Diagnosis of PC, encephalopathies and syndromes with non-progressive chronic neurological involvement, with respiratory complications (Pneumonias or Bronchitis).

Exclusion Criteria:

* Patients affected by immunodeficiency or hemato-oncological process.
* Previous respiratory pathology in itself (not consistent with its underlying pathology)
* Patients with cardiovascular instability.
* Patients with drained pneumothorax.
* Patients with recent pneumonectomy.
* Patients with severe bullae.
* Patients with hemoptysis.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from Quality of Life Related to Health (HRQoL) at 6 month | The PedsQL questionnaires were completed at the beginning of the study, at 6 months after the start of the study.
  It was objectified through a personal interview with the parents, the PedsQL ™ Questionnaire on Pediatric Life Quality in Spanish version was used with the corresponding permission of use. The PedsQL ™ Generic Module investigates four areas or dimensions of the child's HRQoL: Physical, Emotional, Social and School Functioning. To calculate the HRQoL measure, the items were linearly transformed using a five-point Likert scale, on a scale of 0-100.
Change from number of hospitalizations | The number of hospitalizations for respiratory complications that each participant had during the six months before and after the start of the study was recorded.
  Number of admissions due to respiratory complications. It was valued through a personal interview with the parents.

SECONDARY OUTCOMES:
Pulmonary auscultation | It was assessed through study completion, an average of 6 month .
  The presence or absence of adventitious noises was assessed. The conserved vesicular murmur corresponds to normal respiratory noise and indicates good pulmonary ventilation. The adventitious sounds assessed are crackles, wheezing and hypoventilation, indicating poor pulmonary ventilation and bronchial obstruction. The auscultation was assessed using the 3M ™ Littmann® Classic II Pediatric Stethoscope.
Pulsoximetry | It was evaluated through study completion, an average of 6 month .
  It was measured by the finger Pulsioximetro, M-Pulse ™ pediatric.
Heart rate | It was measured through study completion, an average of 6 month.
  It was evaluated using the finger Pulse Oximeter, M-Pulse ™ pediatric
Respiratory Rate | It was measured through study completion, an average of 6 month.
  The number of breathing cycles was valued with the help of a crono for 60 seconds in the rest of the participants, in a noise-free environment.
Sputum | It was measured through study completion, an average of 6 month .
  It was measured in millimeters of secretions with a millimetric glass.
Number of emergency visits | The number of visits to the emergency department due to respiratory complications that each participant had during the six months before and after the study was recorded.
  Number of emergency visits due to respiratory complications. It was valued through a personal interview with the parents.
Number of visits to pediatrician | The number of pediatric visits for respiratory complications that each participant had during the six months before and after of the study was recorded.
  Number of visits to pediatrician due to respiratory complications. It was valued through a personal interview with the parents.

OTHER OUTCOMES:
Thoracic mobility | It was measured through study completion, an average of 6 month.
  The measurement of maximal inspiration, maximal expiration and the difference between both (thoracic expansion) in the sitting position was made using a tape measure marked in increments of 0.1 cm at the level of the fourth intercostal space.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada M Moreno, Doctora, Principal Investigator — Sociedad Española de Cirugía y neumología Torácica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flores JC, Carrillo D, Karzulovic L, Cerda J, Araya G, Matus MS, Llevenes G, Menchaca G, Vargas NA. [Children with special health care needs: prevalence in a pediatric hospital and associated risks]. Rev Med Chil. 2012 Apr;140(4):458-65. doi: 10.4067/S0034-98872012000400006. Spanish. PMID 22854691
- [Background] Marks JH. Pulmonary care of children and adolescents with developmental disabilities. Pediatr Clin North Am. 2008 Dec;55(6):1299-314, viii. doi: 10.1016/j.pcl.2008.08.006. PMID 19041459
- [Background] Schechter MS. Airway clearance applications in infants and children. Respir Care. 2007 Oct;52(10):1382-90; discussion 1390-1. PMID 17894905
- [Background] Hess DR. Airway clearance: physiology, pharmacology, techniques, and practice. Respir Care. 2007 Oct;52(10):1392-6. PMID 17894906
- [Result] Tenenbaum A, Hanna RN, Averbuch D, Wexler ID, Chavkin M, Merrick J. Hospitalization of children with down syndrome. Front Public Health. 2014 Mar 20;2:22. doi: 10.3389/fpubh.2014.00022. eCollection 2014. PMID 24688981
- [Result] Hill CM, Parker RC, Allen P, Paul A, Padoa KA. Sleep quality and respiratory function in children with severe cerebral palsy using night-time postural equipment: a pilot study. Acta Paediatr. 2009 Nov;98(11):1809-14. doi: 10.1111/j.1651-2227.2009.01441.x. Epub 2009 Jul 22. PMID 19627261
- [Result] Littleton SR, Heriza CB, Mullens PA, Moerchen VA, Bjornson K. Effects of positioning on respiratory measures in individuals with cerebral palsy and severe scoliosis. Pediatr Phys Ther. 2011 Summer;23(2):159-69. doi: 10.1097/PEP.0b013e318218e306. PMID 21552079
- [Result] Al-Khaledi B, Lewis M, Maclean JE. Case 2: Recurrent lower respiratory tract infections in a child with Down syndrome. Paediatr Child Health. 2014 Jan;19(1):19-21. doi: 10.1093/pch/19.1.19a. No abstract available. PMID 24627649
- [Result] Kwon YH, Lee HY. Differences of respiratory function in children with spastic diplegic and hemiplegic cerebral palsy, compared with normally developed children. J Pediatr Rehabil Med. 2013;6(2):113-7. doi: 10.3233/PRM-130246. PMID 23803344
- [Result] McCool FD, Rosen MJ. Nonpharmacologic airway clearance therapies: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):250S-259S. doi: 10.1378/chest.129.1_suppl.250S. PMID 16428718
- [Result] Lagerkvist AL, Sten G, Westerberg B, Ericsson-Sagsjo A, Bjure J. Positive expiratory pressure (PEP) treatment in children with multiple severe disabilities. Acta Paediatr. 2005 May;94(5):538-42. doi: 10.1111/j.1651-2227.2005.tb01935.x. PMID 16188740
- [Result] Ortiz Tde A, Forti G, Volpe MS, Carvalho CR, Amato MB, Tucci MR. Experimental study on the efficiency and safety of the manual hyperinflation maneuver as a secretion clearance technique. J Bras Pneumol. 2013 Mar-Apr;39(2):205-13. doi: 10.1590/S1806-37132013000200012. PMID 23670506
- [Result] de Godoy VC, Zanetti NM, Johnston C. Manual hyperinflation in airway clearance in pediatric patients: a systematic review. Rev Bras Ter Intensiva. 2013 Jul-Sep;25(3):258-62. doi: 10.5935/0103-507X.20130043. PMID 24213091
- [Result] Barks L, Shaw P. Wheelchair positioning and breathing in children with cerebral palsy: study methods and lessons learned. Rehabil Nurs. 2011 Jul-Aug;36(4):146-52, 174. doi: 10.1002/j.2048-7940.2011.tb00082.x. PMID 21721395
- [Result] Fitzgerald DA, Follett J, Van Asperen PP. Assessing and managing lung disease and sleep disordered breathing in children with cerebral palsy. Paediatr Respir Rev. 2009 Mar;10(1):18-24. doi: 10.1016/j.prrv.2008.10.003. Epub 2009 Jan 23. PMID 19203740
- See also: Tenenbaum A, Hanna RN, Averbuch D, Wexler ID, Chavkin M, Merrick J. Hospitalization of children with down syndrome. Front Public Health. 2014 Mar 20;2:22. doi: 10.3389/fpubh.2014.00022. eCollection 2014. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3960574/
- See also: Al-Khaledi B, Lewis M, Maclean JE. Case 2: Recurrent lower respiratory tract infections in a child with Down syndrome. Paediatr Child Health. 2014 Jan;19(1):19-21. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3938214/
- See also: Ortiz Tde A, Forti G, Volpe MS, Carvalho CR, Amato MB, Tucci MR. Experimental study on the efficiency and safety of the manual hyperinflation maneuver as a secretion clearance technique. J Bras Pneumol. 2013. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4075822/pdf
- See also: Fitzgerald DA, Follett J, Van Asperen PP. Assessing and managing lung disease and sleep disordered breathing in children with cerebral palsy. Paediatr Respir Rev. 2009 — https://www.clinicalkey.com/#!/content/playContent/1-s2.0-S1526054208000729?returnurl=https:%2F%2Flinkinghub.elsevier.com%2Fretrieve%2Fpii%2FS1526054208000729%3Fshowall%3Dtrue&referrer=https:%2F%2Fwww.ncbi.nlm.nih.gov%2Fpubmed%3Fterm%3DAssessing%2Band%2Bmanaging%2Blung%2Bdisease%2Band%2Bsleep%2Bdisordered%2Bbreathing%2Bin%2Bchildren%2Bwith%2Bcerebral%2Bpalsy%26TransSchema%3Dtitle%26cmd%3Ddetailssearch